CLINICAL TRIAL: NCT00109824
Title: A Phase I Study of Decitabine in Combination With Valproic Acid in Patients With Relapsed/Refractory Non-Hodgkin's Lymphoma
Brief Title: Decitabine With or Without Valproic Acid in Treating Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01465; 0475; CDR0000426523; OSU-0475; NCI-6997; OSU-2004C0119; U01CA076576 (NIH)
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Mantle Cell Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell | interventions — Decitabine; Valproic Acid

ARMS (2):
- Arm I (Experimental): Patients receive decitabine IV over 1 hour on days 1-5 or 1-10. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: pharmacological study; Other: laboratory biomarker analysis
- Arm II (Experimental): Patients receive decitabine as in stage 1 and valproic acid PO TID on days 5-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: decitabine; Drug: valproic acid; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: decitabine — Given IV
  Other Names: 5-aza-dCyd; 5AZA; DAC
  Arms: Arm II
Drug: valproic acid — Given PO
  Other Names: Alti-Valproic; Depakene; Novo-Valproic; VA
  Arms: Arm II
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Drugs used in chemotherapy, such as decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Valproic acid may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving decitabine together with valproic acid may be an effective treatment for non-Hodgkin's lymphoma. This phase I trial is studying the side effects and best dose of decitabine and valproic acid in treating patients with relapsed or refractory aggressive B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the minimally effective pharmacological dose (MEPD) of single-agent decitabine in patients with relapsed or refractory aggressive B-cell non-Hodgkin's lymphoma.

II. Determine the maximum tolerated dose of valproic acid when administered with the MEPD of decitabine in these patients.

III. Determine the MEPD of valproic acid when administered with decitabine in these patients.

IV. Determine the toxic effects of decitabine alone and in combination with valproic acid in these patients.

SECONDARY OBJECTIVES:

I. Determine the response rate in patients treated with these drugs. II. Determine the pharmacokinetics of these drugs in these patients.

OUTLINE: This is a dose-escalation study. Patients are assigned to 1 of 2 treatment stages.

STAGE 1: Patients receive decitabine IV over 1 hour on days 1-5 or 1-10. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

STAGE 2: Patients receive decitabine as in stage 1 and valproic acid orally (PO) thrice daily (TID) on days 5-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

For both stages, patients who achieve an objective response (complete response [CR], unconfirmed CR, or partial response) may discontinue study treatment and undergo stem cell transplantation, if eligible.

PROJECTED ACCRUAL: Approximately 18-42 patients (18 for stage 1 and 24 for stage 2) will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed aggressive B-cell non-Hodgkin's lymphoma (NHL), including any of the following subtypes:

  * Mantle cell lymphoma
  * Diffuse large cell lymphoma
  * Burkitt's lymphoma
  * Transformed NHL* arising from a previously diagnosed low-grade lymphoma, including any of the following:

    * Follicular lymphoma
    * Small lymphocytic lymphoma
    * Chronic lymphocytic leukemia
* Relapsed or refractory disease

  * Relapsed or refractory disease must have occurred during the most recent prior therapy
* Has accessible tissue for biopsy OR evidence of ≥ 50% bone marrow involvement AND willing to undergo serial biopsy
* Not eligible for OR refused curative stem cell transplantation
* No active or untreated CNS lymphoma
* Performance status - ECOG 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 75,000/mm^3
* AST and ALT ≤ 2.5 times upper limit of normal
* Bilirubin ≤ 1.5 mg/dL
* Creatinine ≤ 2.0 mg/dL
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known HIV positivity
* No ongoing or active infection
* No other uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance
* Prior stem cell transplantation allowed
* Recovered from all prior biologic therapy-related toxicity
* Recovered from all prior chemotherapy-related toxicity
* No other concurrent chemotherapy unless it is used in the chronic daily setting for other medical conditions, including pulmonary, rheumatologic, or adrenal disorders
* No concurrent corticosteroids unless they are used in the chronic daily setting for other medical conditions, including pulmonary, rheumatologic, or adrenal disorders
* Recovered from all prior radiotherapy-related toxicity
* No concurrent palliative radiotherapy
* Recovered from all prior therapy-related toxicity
* No concurrent anticonvulsants, including valproic acid (except as used in this study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-03; Primary Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
MEPD of single agent decitabine defined as the dose where an 80% decrease in DNMT1 protein level and a 100% increase in re-expression of the methylated target genes are noted in 5 of 6 patients, with DLT in less than or equal to 1 patient | 28 days
MTD of valproic acid in combination with the MEPD of decitabine defined as the dose level below that dose at which greater than or equal to 2 DLT are observed and that results in less than or equal to 1 DLT in 6 patients using CTCAE v3.0 | 28 days
MEPD of valproic acid and decitabine defined as the dose where an 80% decrease in DNMT1 protein level and a 100% increase in re-expression of the methylated target genes are noted in 5 of 6 patients, with DLT in less than or equal to 1 patient | 28 days
Toxicities of single agent decitabine alone and in combination with valproic acid assessed using CTCAE v3.0 | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kristie Blum, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States